CLINICAL TRIAL: NCT00886535
Title: An Observational Trial of the Effect of Pharmacogenomics Differences in Phase I and II Metabolism of Tamoxifen on Efficacy and Toxicity
Brief Title: Effect of Pharmacogenomics Differences in Phase I and II Metabolism of Tamoxifen on Efficacy and Toxicity
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Leah Cream, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Other Study IDs: PSHCI 08-047
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
Keywords: breast cancer; hot flashes; tamoxifen
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Hot Flashes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will be an open-label prospective observational trial designed to test associations between polymorphisms of candidate genes and tamoxifen. Pre- and post-menopausal women taking tamoxifen as standard therapy or chemopreventive therapy will be included in this study.

DETAILED DESCRIPTION:
This study will be an open-label prospective observational trial designed to test associations between polymorphisms of candidate genes (focusing initially on the UGT2B7 enzyme) and tamoxifen (TAM) toxicity. Pre- & post-menopausal women (aged ≥18 years) taking TAM (20 mg/day) as standard therapy or chemopreventive therapy will be included in this study. Patients will be enrolled after they complete all primary surgery, radiation, and adjuvant chemotherapy. Patients will be excluded if they are undergoing other adjuvant endocrine therapies. Other reasons for exclusion will include patients who are pregnant or lactating, or are currently on corticosteroids, phenobarbital, or megestrol acetate. The goal will be to recruit a total of 45 eligible patients over a 1 year accrual period. The investigators expect to treat ~50 new patients per year with TAM at the standard dose of 20 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving tamoxifen for adjuvant therapy of breast cancer or ductal carcinoma in situ, or as chemoprevention
* Age 18 years and above
* May be pre- and post-menopausal
* Females
* Patients may be at any point in their hormonal treatment, but must have completed any planned surgery, radiation and chemotherapy
* Must use a reliable form of birth control

Exclusion Criteria:

* Pregnant
* Breastfeeding
* Concurrent use of corticosteroids, megestrol, or phenobarbital
* History of allergy to tamoxifen
* Unwilling to have a yearly gynecological exam

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females, age 18 years of age and above. Patients receiving tamoxifen for adjuvant therapy of breast cancer or ductal carcinoma in situ or as chemoprevention.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Hot flashes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leah Cream, MD, Principal Investigator — Penn State Hershey Cancer Institute
Locations (1):
- Penn State Hershey Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
After determining if data is valuable